CLINICAL TRIAL: NCT05666635
Title: A Phase I Clinical Trial to Assess the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of LTC004 in Patients With Advanced or Metastatic Malignancies
Brief Title: Study of LTC004 in Subjects With Advanced Malignant Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Letolab (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: LTC004-101
Record Dates: First submitted 2022-11-10; First posted 2022-12-28 (Actual); Last update posted 2022-12-28 (Actual); Status verified 2022-12

CONDITIONS: Adult Solid Tumor

STUDY DESIGN:
Intervention Model Description: Participants will be assigned to sequentially escalating dose cohorts of LTC004
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental：LTC004 (Experimental): Monotherapy, dose escalation
  Interventions: Biological: LTC004

INTERVENTIONS:
Biological: LTC004 — LTC004 Phase I:Participants will be allocated to one of the following dose groups: 3, 15, 45, 90, 180，270,360 and 450 ug/kg, and receive a treatment of LTC004 followed by 21 days of dose limited toxicity (DLT) observation period.
  Phase Ib indication exploration
  Other Name: LTC004 for Injection

SUMMARY:
This was a multicenter, open, multi-cohort PHASE I study, consisting of 2 phases: Phase Ia (Phase Ia dose escalation) and Phase Ib (Phase Ib multi-cohort expansion). The objective of this study was to evaluate safety, tolerability, pharmacokinetic， Pharmacodynamics and biological characteristics, and initial efficacy in advanced malignant tumors.

DETAILED DESCRIPTION:
Phase I dose escalation phase：This study predicted a total of 8 dose groups, 3, 15, 45, 90, 180，270，360 and 450 ug/kg.

Phase Ib expansion phase: This phase is the multi-cohort indication expansion phase. Based on the data obtained in phase I, chose an appropriate dose continue to explore multi-cohort indications.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged 18 to 75 years (including upper and lower limit) at the time of signing the informed consent form (ICF)；
2. Subjects with locally advanced or metastatic solid tumors or lymphoma who have histologically or cytologically confirmed inoperable disease at screening and have failed from standard treatment，or cannot tolerate standard treatment and/or currently have no effective standard treatment；
3. Patients must have at least 1 lesion that qualifies as a target lesion；
4. ECOG≤1；
5. Life expectancy ≥3 months；
6. Adequate organ function；
7. Patients who have received any chemotherapy or anti-tumor monoclonal antibody drugs within 4 weeks prior to the first dose of study drug (excluding mitomycin and nitrosoureas within 6 weeks prior to the first dose of study drug）; small molecule targeted drugs within 2 weeks prior to the first dose of study drug; Chinese medicine therapy (Chinese medicine therapy with clear anti-tumor indications in the package insert ）within 4 weeks prior to the first dose of study drug；
8. Patients, both females and males, of reproductive potential must agree to use adequate contraception during and for 6 months after the last infusion of LTC004.
9. Understands and provides written informed consent and willing to follow the requirements specified in protocol

Exclusion Criteria:

1. History of severe hypersensitivity reactions to other mAbs.
2. Untreated, unstable or uncontrolled central nervous system (CNS) metastases with following exceptions:A. Clinically stable MRI scans (at least 2 consecutive scans within prior 6 months including 1 scan within 28 days prior to screening) and no progressive or uncontrolled neurologic symptoms or signs (e.g., seizures, headaches, central nausea/emesis, progressive neurologic deficits, papilledema) for at least 4 weeks prior to the first study treatment;
3. Patients with uncontrolled pleural effusion, pericardial effusion or abdominal effusion (requiring repeated drainage, more than one month or more frequently) as judged by the investigator at screening;
4. Patients with untreated or clinically uncontrolled spinal cord compression (except for those who have been treated and have stable symptoms and image for at least 4 weeks before the first dose, and no evidence of cerebral edema, and no need for glucocorticoid therapy);
5. Concurrent malignancy within 5 years prior to entry, except for adequately treated cervical carcinoma-in-situ, localized squamous cell cancer of the skin, basal cell carcinoma;
6. Moderate to severe dyspnea at rest, severe primary lung disease required for continuous oxygen therapy, or clinically active interstitial lung disease (ILD) or pneumonia due to advanced cancer or its complications; ≥ Grade 3 interstitial pneumonia during previous anti-tumor treatment;
7. History of moderate to severe dyspnea at rest due to advanced cancer or their complications, severe primary lung disease, current need of continuous oxygen therapy, or clinically active interstitial lung disease (ILD) or pneumonitis.
8. Severe infection within 4 weeks before the first dose, including but not limited to bacteremia requiring hospitalization, severe pneumonia, etc.; active infection with CTCAE ≥ grade 2 requiring systemic antibiotics within 2 weeks before the first dose；
9. History of serious cardiovascular and cerebrovascular diseases, including but not limited to: severe heart rhythm or conduction abnormalities, such as ventricular arrhythmia requiring clinical intervention, II-III degree atrioventricular block, etc.; acute coronary syndrome, congestive heart failure, aortic dissection, stroke or other grade 3 and above cardiovascular and cerebrovascular events within 6 months before the first dose; New York Heart Association (NYHA) functional classification ≥ II or left ventricular ejection fraction (LVEF) < 50% or clinically uncontrolled hypertension (systolic blood pressure ≥ 160 mmHg and/or diastolic blood pressure ≥ 100 mmHg);
10. Patients who have any known liver disease, including chronic hepatitis B (HBsAg positive and HBV DNA ≥ ULN of local site and excluding hepatitis caused by drugs or other reasons), hepatitis C, autoimmune hepatic disorders, primary biliary cirrhosis or sclerosing cholangitis; Patients who have concurrent, serious, uncontrolled infections or known infection with HIV, or have a diagnosed acquired immunodeficiency syndrome (AIDS); or an uncontrolled autoimmune disease, or have undergone organ transplant；
11. Syphilis positive patients at screening；
12. Patients with active autoimmune diseases (such as systemic lupus erythematosus, rheumatoid arthritis, vasculitis, etc.) at screening, or have suffered from autoimmune diseases that may relapse, except for patients with clinically stable autoimmune thyroid disease；
13. History of immunodeficiency disease , including positive human immunodeficiency virus (HIV) serum test；
14. Patients who have experienced bleeding symptoms of significant clinical significance within 3 months before the first dose; Subjects who had a significant cough of blood and hemoptysis of half a teaspoon (2.5 mL) or more per occasion within 4 weeks prior to the first dose of study drug; arterial/venous thrombotic events such as cerebrovascular accident, deep venous thrombosis, pulmonary embolism within 6 months prior to the first dose; and those who were receiving anticoagulant therapy at screening；
15. Patients who have received systemic immunosuppressive therapy (including but not limited to glucocorticoids, cyclophosphamide, azathioprine, methotrexate, thalidomide, etc.) within 2 weeks before the first dose；
16. Immunomodulatory drugs within 2 weeks (or 5 drug half-lives, whichever is longer) before the first dose, including but not limited to thymosin, IL-2, IL-15, interferon, etc.
17. Receiving non-thoracic radical radiotherapy > 30 Gy within 4 weeks before the first dose, thoracic radiotherapy > 30 Gy within 24 weeks before the first dose, and palliative radiotherapy ≤ 30 Gy within 14 days before the first dose.
18. Received other unmarketed clinical study drugs or treatments within 4 weeks before the first dose.
19. Use of live or attenuated vaccines within 4 weeks prior to the first dose, or anticipated need for live or attenuated vaccines during the study.

20:Received major surgery within 4 weeks prior to the first dose (except for procedures for diagnostic purposes), anticipated major surgery during the study (except for procedures for diagnostic purposes), or diagnostic or less invasive surgery within 7 days prior to the first dose (not in this range for needle biopsy).

21：Have not recovered from previous anti-tumor treatment， CTCAE 5.0 grade evaluation ≤ 1 (alopecia and grade 2 neurotoxicity caused by chemotherapeutic drugs, as well as grade 2 hypothyroidism caused by anti-tumor treatment); 22：Patients who have previously received allogeneic bone marrow/hematopoietic stem cell transplantation or solid organ transplantation.

23：Pregnant and lactating women. 24：The subjects have a history of other serious systemic diseases or any other reason (patients with mental illness, alcoholism, drug abuse or drug abuse that may affect the compliance of the trial) should not participate in this trial as judged by investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 368 (Estimated)
Dates: Start 2022-12 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Adverse Event (AE) | up to 12 months
  safety and tolerability as measured by the incidence of treatment-emergent adverse events.
Number of participants with DLTs | up to 21 days
  DLTs as measured by the incidence during Cycle 1.

SECONDARY OUTCOMES:
Objective response rate (ORR) | up to 12 months
  The ORR is defined as the proportion of subjects with confirmed CR or confirmed PR, based on RECIST Version 1.1.
Serum concentrations of LTC004 | up to 12 months
  Concentration data will be summarized by dose level
Immunogenicity of LTC004 | up to 12 months
  Results will be summarized by dose level
Serum concentrations of cytokines and T cell | up to 12 months
  including IFNγ, TNF-α, IL-1B, IL-6, IL-10，total T cells, CD8+ T cells, NK cells and Treg cells